CLINICAL TRIAL: NCT01728064
Title: Safety and Efficacy Study of EPI-743 on Visual Function in Patients With Friedreich's Ataxia
Brief Title: Safety and Efficacy of EPI-743 in Patients With Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPI2010-006
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's; Ataxia; FRDA; FA; EPI-743; Edison
MeSH Terms: conditions — Friedreich Ataxia; Ataxia | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo capsules three times daily
  Interventions: Drug: Placebo
- EPI-743 400 mg (Active Comparator): EPI-743 at a dose of 400 mg three times daily
  Interventions: Drug: EPI-743 400 mg
- EPI-743 200 mg (Active Comparator): EPI-743 at a dose of 200 mg three times daily
  Interventions: Drug: EPI-743 200 mg

INTERVENTIONS:
Drug: Placebo — Placebo capsules
  Arms: Placebo
Drug: EPI-743 400 mg
  Arms: EPI-743 400 mg
Drug: EPI-743 200 mg
  Arms: EPI-743 200 mg

SUMMARY:
The purpose of this study is to examine the effects of EPI-743 on visual function and neurologic function in patients with Friedreich's ataxia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of genetically confirmed Friedreich's ataxia
2. Visual acuity at baseline more than 15 letters on EDTRS at four meters
3. FARS score of 20 to 90
4. Agreement to use contraception if within reproductive years (see specifics in section D1, page 21)
5. Hormone replacement therapy, if used, must remain stable for the duration of the study
6. Willingness and ability to comply with study procedures
7. Willingness and ability to arrive at study site day prior to evaluations
8. Abstention from use of dietary supplements and non-prescribed medications at least 30 days prior to initiation of treatment and for the duration of the study. This would specifically include idebenone, Coenzyme Q10 and vitamin E
9. Abstention from use of other investigative or non-approved drugs within 30 days of enrollment and for the duration of the study

Exclusion Criteria:

1. Allergy to EPI-743 or sesame oil or nuts
2. Clinically significant bleeding condition or abnormal PT/PTT INR (INR > two; PTT > two-times normal)
3. Liver insufficiency with LFTs greater than three-times upper normal limit at screening
4. Renal insufficiency with creatinine > 1.5 at screening
5. Fat malabsorption syndromes
6. Any other respiratory chain diseases of the mitochondria or inborn errors of metabolism
7. Any other ophthalmologic conditions
8. History of alcohol or drug abuse
9. Clinically significant cardiomyopathy with ejection fraction < 40 percent at screening
10. Clinically significant arrhythmia within past two years requiring treatment
11. Anticoagulant therapy within 30 days of enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12-31 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Visual Function
  Low contrast visual acuity

SECONDARY OUTCOMES:
Color vision
  Roth 28 hue test
Neurologic function
  Friedreich's ataxia rating scale
Neuromuscular function
  25-foot walk test
Neuromuscular function
  9-hole peg test
Quality of life
  SF-36
Disease biomarkers
  Blood biomarker levels
Cardiac function
  Echocardiogram
Safety
  Number of adverse events
Disease improvement
  Patient Global Improvement Scale
Visual Function | Baseline, Months 3, 6, 9 and 12
  Visual field exam

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Edison Pharmaceuticals Web Site — http://edisonpharma.com